CLINICAL TRIAL: NCT03720210
Title: Pilot Study for Treatment of Amiodarone-Induced Thyroiditis With Radiofrequency Ablation
Brief Title: Radiofrequency Ablation for Amiodarone-induced Thyrotoxicosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very low enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marius Stan, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-004450
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Results first posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Amiodarone-Induced Thyrotoxicosis
Keywords: Hyperthyroidism; RFA
MeSH Terms: conditions — Hyperthyroidism

STUDY DESIGN:
Intervention Model Description: Open label single interventional series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- RFA group (Experimental): RFA
  Interventions: Device: RFA

INTERVENTIONS:
Device: RFA — Radiofrequency ablation of a portion of thyroid parenchyma to treat amiodarone-induced thyrotoxicosis

SUMMARY:
Investigators intend to study the changes in thyroid hormone storage and production in amiodarone-induced thyrotoxicosis patients after RFA therapy.

DETAILED DESCRIPTION:
Investigators plan to identify patients with amiodarone-induced thyrotoxicosis (AIT) that failed to respond to medical therapy or have developed side effects from medical therapy or are considered high risk for such therapy.

These patients will be offered the option to undergo radiofrequency ablation (RFA) of a portion of the thyroid gland in order to decrease thyroid hormone production and/or to inactive the existing thyroid hormone store before their leakage into the circulation.

Investigators will follow these patients to assess their clinical response as well as their thyroid values. The safety of the procedure will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Are adults
* Have overt thyrotoxicosis (within 2 weeks prior to enrollment)
* Are receiving medical therapy for AIT
* Are able to understand the study procedures and to comply with them for the entire length of the study
* Have not normalized their thyroid levels after one month of standard therapy or
* Have persistent and clinically significant thyrotoxicosis (less than 25% decrease in T4 value or patients requiring hospitalization with Congestive heart failure (CHF), tachyarrhythmias, hemodynamic instability or similar co-morbidities) after 2 weeks of standard therapy where additional medical therapy is deemed unlikely to be beneficial or with high risk of side-effects (e.g. hepatotoxicity of antithyroid medications, agranulocytosis of potassium perchlorate or ATD or fluid retention associated with steroids).

Exclusion Criteria:

* Pregnancy
* Patients with prior neck surgery or neck radiation
* Patients with neck anatomy that precludes easy access by RFA to the entirety of thyroid parenchyma
* Patients on anticoagulation therapy
* Patients with comorbidities deemed too high of a risk for general anesthesia
* Treatment with another investigational drug or intervention (within 6 weeks of planned RFA).
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius N Stan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- RFA Group: RFA (Radiofrequency Ablation)
  RFA: Radiofrequency ablation of a portion of thyroid parenchyma to treat amiodarone-induced thyrotoxicosis
Period: Overall Study
Arm/Group | RFA Group
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | RFA Group
Number analyzed (Participants) | 1
Age, Customized [Count of Participants; unit: Participants]
  Age 31 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Free T4 Response Post RFA
Description: Thyroid tests
Time Frame: 3 - 6 months
Population: The one subject enrolled did not return for follow up. Data not collected or analyzed.
Arm/Group | RFA Group
Number analyzed (Participants) | 0

2. Primary Outcome: Total T3 Response Post RFA
Description: Thyroid tests
Time Frame: 3 - 6 months
Population: The one subject enrolled did not return for follow up. Data not collected or analyzed.
Arm/Group | RFA Group
Number analyzed (Participants) | 0

3. Secondary Outcome: Pain Related to RFA Procedure
Description: McGill Pain Questionnaire
Time Frame: 1 - 2 months
Population: The one subject enrolled did not return for follow up. Data not collected or analyzed.
Arm/Group | RFA Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Thyroid-stimulating Hormone (TSH) Response Post RFA
Description: Thyroid tests
Time Frame: 3 - 6 months
Population: The one subject enrolled did not return for follow up. Data not collected or analyzed.
Arm/Group | RFA Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from RFA procedure to 72 hours post RFA procedure.
Arm/Group | RFA Group
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Lack of interested & suitable candidates. The one subject enrolled was lost to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03720210/Prot_SAP_000.pdf